CLINICAL TRIAL: NCT00686985
Title: A Phase II Study of Docetaxel - Carboplatin As Second Line Treatment in Patients with Refractory or Relapsed Small Cell Lung Cancer
Brief Title: Docetaxel - Carboplatin As Second Line Treatment in Patients with Small Cell Lung Cancer
Acronym: DOCAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. B. Biesma (Other)
Responsible Party: Sponsor-Investigator, Dr. B. Biesma, MD, PhD, Pulmonologist, Jeroen Bosch Ziekenhuis
Organization: Jeroen Bosch Ziekenhuis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOCAR study
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2024-09-20 (Actual); Status verified 2024-03

CONDITIONS: Small Cell Lung Cancer
Keywords: Docetaxel; Carboplatin; chemotherapy; relapse SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Carboplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Carboplatin, docetaxel

INTERVENTIONS:
Drug: Carboplatin, docetaxel — Carboplatin AUC 5, Docetaxel 75 mg/m2, q 3 weeks, 4-6 cycles, 12-18 weeks

SUMMARY:
Phase II studies with docetaxel in first line - and second line treatment of SCLC demonstrated that docetaxel is an active agent in these patient groups. Therefore docetaxel seems suitable for evaluation in combination with other cytotoxic drugs active in this disease. A phase II study in previously untreated patients with SCLC shows that the combination docetaxel and cisplatin/carboplatin is an active and well tolerated regimen in extensive SCLC.

DETAILED DESCRIPTION:
Background:

Small cell lung cancer (SCLC) is diagnosed in approximately 15 % of all the lung cancer cases. SCLC is recognized by its rapid tumor growth, with a high chemo- and radio sensitivity, and by its high metastasizing potential. Patients with extensive-stage disease have a 5-year survival rate of 1% to 2%.

Almost 2/3 of the patients have already extensive disease (ED) upon diagnosis.The recommended treatment of ED-SCLC is systemic chemotherapy, considered to be the standard first line treatment option in all patients with SCLC regardless of performance status and age. World-wide, the most commonly used regimen for 1st line treatment is the combination of cisplatin-etoposide, while in the Netherlands the cyclophosphamide, doxorubicin and etoposide regimen is widely used.Survival outcome with these regimens appear similar.

Unfortunately, relapses occur in all patients and responses to second-line chemotherapy have proven to be of short term. Until recently, there were no registered drugs for treatment of relapsing SCLC. Phase II studies with docetaxel in first line - and second line treatment of SCLC demonstrated that docetaxel is an active agent in these patient groups. Therefore docetaxel seems suitable for evaluation in combination with other cytotoxic drugs active in this disease. Until now no studies have been performed with a combination of docetaxel and platinum in this group of previously treated SCLC patients.

A phase II study in previously untreated patients with SCLC shows that the combination docetaxel and cisplatin/carboplatin is an active and well tolerated regimen in extensive SCLC.

Study objectives:

To evaluate the anti-tumor activity of a docetaxel/carboplatin regimen in patients with refractory or relapsed SCLC. Furthermore to asses the safety profile of the docetaxel/carboplatin combination.

Trial design:

This study will be a open label non-randomized study conducted in patients with refractory or relapsed SCLC. It is a phase II study with 50 patients.

Docetaxel infusion 75 mg/m2, carboplatin AUC = 6 mg/ml·min day 1, every 21 days for 4-6 cycles.

Population:

Patients with histologically or cytologically proven SCLC at the first diagnosis with refractory or relapsed SCLC after first line treatment. Signed informed consent. Age > 18 years. WHO ps 0,1 or 2.

Endpoints:

Primary endpoint: response rate. Secondary endpoint(s): time to progression, response duration, safety profile and survival.

Stress and risks for the patient:

Hospital visits and tests are not different from the standard treatment. Stress due to adverse events is not essential higher estimated. Special risks are not expected. Frequently medical examination and control of laboratory results will be done. Detailed instruction will be given about what do to in case of serious toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven SCLC at the first diagnosis
* Refractory or relapsed SCLC
* Measurable disease according to RECIST criteria
* There must be a minimum of 2 weeks between the end of prior radiotherapy and study entry. (No more than 30% of available bone marrow should have been irradiated as recommended by the RTOG).
* Patients must have fully recovered from toxic effects of previous antitumor therapy.
* Age > 18 years.
* WHO performance status 0- 2 (Appendix II).
* Hb > 6.0 mmol/L,

  * Neutrophils > 1.5 x 109/L,
  * Platelets > 100 x 109/L·
* Total bilirubin < the upper-normal limits of the institutional normal values.
* ALAT (SGPT), ASAT (SGOT) < 2.5 times the upper-normal limits of the institutional normal values.
* Alkaline Phosphatase < 5 times the upper-normal limits of the institutional normal values. If AP > 2.5 x ULN then ALAT and ASAT must be <1.5 x ULN, otherwise, the patient is not eligible
* Creatinine < 140 mmol/L; or creatinine clearance according to Cockcroft formula >50 ml/min·
* Signed informed consent prior to beginning protocol specific procedures

Exclusion Criteria:

* More than one line of chemotherapy for metastatic disease
* Treatment with a platinum compound during the last 3 months before randomisation
* Pregnant or lactating women or women of childbearing potential not adhering to adequate anticonceptive measures
* Evidence of (other) active invasive malignancy other than non-melanoma skin cancer.
* Clinical evidence CNS metastases.
* Symptomatic peripheral neuropathy > grade 2 according (NCI CTC, Appendix III)Definite contraindications for the use of corticosteroids
* Concurrent treatment with other experimental drugs.
* Participation in another clinical trial with any investigational drug within 30 days prior to study screening.
* Concurrent treatment with any other cytotoxic anti-cancer therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Response rate | 2 yrs

SECONDARY OUTCOMES:
Time to progression; Response duration; Survival; Safety profile | 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: B Biesma, Dr., Principal Investigator — Jeroen Bosch Ziekenhuis
Locations (1):
- B. Biesma, 's-Hertogenbosch, North Brabant, Netherlands